CLINICAL TRIAL: NCT03181334
Title: The C-SPAN Coalition: Colorectal Cancer Screening and Patient Navigation
Acronym: C-SPAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other); John Peter Smith Health Network (Unknown)
Responsible Party: Principal Investigator, Keith Argenbright, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU 012016-034
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Cancer
Keywords: colorectal; cancer; neoplasm; CRC screening; FIT; Fecal Immunochemical Test
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Branch I (Active Comparator): Condition 1: (Standard Intervention)
  Mailed fecal immunochemical test (FIT) kit including the following:
  Invitation letter to complete free colorectal cancer (CRC) screening.
  Interventions: Behavioral: Branch I
- Branch II and Branch III (Experimental): Condition 2: (Time Guideline)
  Mailed fecal immunochemical test (FIT) kit including the following:
  Invitation to complete free colorectal cancer (CRC) screening within a specified time frame:
  Branch II - Brief Time (1-week)
  Branch III - Extended Time (3-weeks)
  Interventions: Behavioral: Branch II; Behavioral: Branch III
- Branch IV and Branch V (Experimental): Condition 3: (Time Guideline + Incentive)
  Mailed fecal immunochemical test (FIT) kit including the following:
  Invitation to complete free colorectal (CRC) screening within a specified time frame with a monetary incentive:
  Branch IV - High Incentive
  Branch V - Low Incentive
  Interventions: Behavioral: Branch IV; Behavioral: Branch V

INTERVENTIONS:
Behavioral: Branch I — FIT kits and a Standard (control) invitation letter to complete CRC screening is mailed to the homes of eligible patients.
  Other Names: Condition 1 - Standard Intervention
  Arms: Branch I
Behavioral: Branch II — FIT kits and a Brief Time invitation to complete CRC screening is mailed to the homes of eligible patients. Time letters are used to evaluate the effect of procrastination on CRC screening compliance.
  Participants are assigned to the following intervention:
  Branch II: Invitation letter to participate in free CRC screening, requesting they return the kit within 1-week.
  Other Names: Condition 2 - Time Guideline; Brief Time
  Arms: Branch II and Branch III
Behavioral: Branch III — FIT kits and an Extended Time invitation to complete CRC screening is mailed to the homes of eligible patients. Time letters are used to evaluate the effect of procrastination on CRC screening compliance.
  Participants are assigned to the following intervention:
  Branch III: Invitation letter to participate in free CRC screening, requesting they return the kit within 3-weeks.
  Other Names: Condition 2 - Time Guideline; Extended Time
  Arms: Branch II and Branch III
Behavioral: Branch IV — FIT kits and a Time + Incentive invitation to complete CRC screening is mailed to the homes of eligible patients. Time + Incentive letters are used to evaluate the effect of incentive on procrastination in CRC screening compliance.
  Participants are assigned to the following intervention:
  Branch IV: Invitation letter to participate in free CRC screening, requesting they return the kit within 1-week for a "higher" incentive or within 3-weeks for a "lower" (half of the higher) incentive.
  Other Names: Condition 3 - Time Guideline + Incentive; High Incentive
  Arms: Branch IV and Branch V
Behavioral: Branch V — FIT kits and a Time + Incentive invitation to complete CRC screening is mailed to the homes of eligible patients. Time + Incentive letters are used to evaluate the effect of incentive on procrastination in CRC screening compliance.
  Participants are assigned to the following intervention:
  Branch V: Invitation letter to participate in free CRC screening, requesting they return the kit within 1-week for a "higher" (same as lower Branch IV) or within 3-weeks for a "lower" (half of lower Branch IV) incentive.
  Other Names: Condition 3 - Time Guideline + Incentive; Low Incentive
  Arms: Branch IV and Branch V

SUMMARY:
Participants will be mailed an invitation to complete CRC screening along with a fecal immunochemical test (FIT) kit, containing a 1-sample "Polymedco Over the Counter (OC) Sensor FIT", simplified English/Spanish instructions on performing the test, educational information about colorectal cancer screening and a return mailer with prepaid postage.

Processes that will be used to promote screening completion include automated and "live" phone call reminders to encourage completion of FIT testing.

Participants will be randomly assigned to 1 of 5 interventions across 3 conditions, described below:

1. Condition 1 (Standard Intervention):

   * Branch I: Participants assigned to the control condition will receive a FIT kit and the standard invitation letter to participate in free screening.
2. Condition 2 (Time Guideline):

   * Branch II: Participants will receive a FIT kit and invitation letter to participate in free screening with a 1-week time restriction.
   * Branch III: Participants will receive a FIT kit and invitation letter to participate in free screening with a 3-week time restriction.
3. Condition 3 (Time Guideline + Incentive):

   * Branch IV: Participants will receive a FIT kit and invitation letter to participate in free screening requesting they return the kit within 1-week for a "higher" monetary incentive or within 3 weeks for a "lower" (half of the higher) monetary incentive.
   * Branch V: Participants will receive a FIT kit and invitation letter to participate in free screening requesting they return the kit within 1-week for a "higher" (same as lower in Branch IV) monetary incentive or within 3 weeks for a "lower" (half of the higher) monetary incentive.

Participants with a normal test result will receive a personal letter confirming this with invitations to complete a repeat screening in subsequent year(s). Participants receiving an abnormal FIT result will be navigated to complete a diagnostic colonoscopy.

Participants continuing in the screening program in subsequent years will receive letters emphasizing the importance of repeat screening to prevent adverse CRC outcomes.

DETAILED DESCRIPTION:
Eligible subjects will be identified from John Peter Smith (JPS) Health Network. A preliminary aggregate report suggests 10,000 patients may be identified for screening evaluation.

Data compilation and management will be centralized at the University of Texas (UT) Southwestern Medical Center - Moncrief Cancer Institute (MCI) using John Peter Smith Health Network administrative claims data to assess screening rates while individually identifying patients not up-to-date with screening. Data will be queried to identify all 50-74 year olds who are potentially eligible for program inclusion.

Data sources will include:

1. The existing database of John Peter Smith patients who are part of a previous CRC screening study (STU 082012-086)
2. Administrative and electronic medical record databases from JPS

Patient datasets provided by John Peter Smith Health Network will be obtained through a data use agreement. Inclusion/exclusion criteria will be applied prior to data transfer. The dataset will be transferred through secure, data encrypted transfer systems data encrypted universal serial bus (USB) drives.

Data required for inviting patients to screening and follow-up provided by JPS will be imported into the study tracking database. The tracking database facilitates the day to day program activities and associated data collection, maintaining work lists of patients who have been mailed fecal immunochemical test (FIT) kits and are due for a follow up phone reminder to complete and return the test. The database also accepts updated patient results, such as FIT and colonoscopy test results.

Procedures:

The screening outreach team will be responsible for sending out all invitation letters, tracking results, and facilitating follow up for patients with normal and abnormal FIT tests. Included with the invitation letter, will be a FIT kit, containing a 1-sample Polymedco OC Sensor FIT, simplified English/Spanish instructions on performing the test, educational information about CRC screening and a return mailer with prepaid postage. Completing the test will not require any dietary or medication restrictions for the patient.

Screen eligible individuals will be randomized to 1 of 5 study interventions across 3 conditions (arms) and mailed the appropriate screening invitation letter as described below.

1. Condition 1 (Standard Intervention):

   * Branch I: Participants assigned to the control condition will receive a FIT kit and the standard invitation letter to participate in free screening.
2. Condition 2 (Time Guideline):

   * Branch II: Participants will receive a FIT kit and invitation letter to participate in free screening with a request that they complete the test and mail back within 1-week.
   * Branch III: Participants will receive a FIT kit and invitation letter to participate in free screening with a request that they complete the test and mail back within 3-weeks.
3. Condition 3 (Time Guideline + Incentive):

   * Branch IV: Participants will receive a FIT kit and invitation letter to participate in free screening requesting that they complete the test and mail back within 1-week for a "higher" monetary incentive or within 3 weeks for a "lower" (half of the higher) monetary incentive.
   * Branch V: Participants will receive a FIT kit and invitation letter to participate in free screening requesting that they complete the test and mail back within 1-week for a "higher" (same as lower in Branch IV) or within 3 weeks for a "lower" (half of the higher) monetary incentive.

Patients invited to participate in screening will receive automated telephone calls at the time of invitation. "Live" reminder phone calls will begin at three weeks post invitation for those patients not yet returning a test kit. Bilingual (English/Spanish) program staff will use standardized scripts when completing these calls.

Patients receiving a normal test result will receive a personal letter confirming this with invitations to complete a repeat screening in subsequent year(s).

Patients receiving an abnormal FIT result will be navigated to complete a diagnostic colonoscopy in the Endoscopy suite at JPS hospital. These patients will be contacted by the screening team to be scheduled for pre-operative appointment, after which the patient will then be scheduled for a colonoscopy. The study team's goal will be to schedule and complete colonoscopies within 8 weeks of the abnormal FIT result. If a patient prefers to schedule their colonoscopy with a Non-JPS primary care physician or provider, they will be allowed to do so. In such circumstances the study team will navigate patients to colonoscopy and follow-up with their own provider as with all other JPS patients.

All results and recommendations will also be communicated with both the patient and primary care provider via mail within one week of receiving the result.

Patients identified with colorectal cancer will be navigated to a treatment consultation visit with a surgical or medical oncology clinic, if the diagnosing colonoscopist has not already scheduled this follow-up appointment. The study team's goal will be for patients to be scheduled for this first consultation visit within one week of the CRC diagnosis. Patients will receive reminder phone calls for these visits at both five days and two days prior to the scheduled appointment.

ELIGIBILITY:
Inclusion Criteria:

* Uninsured or Underinsured
* English or Spanish speaking
* No history of colon cancer or colon resection
* No history of inflammatory bowel disease
* Colonoscopy not completed in the last 10 years
* Sigmoidoscopy not completed in the last 5 years
* Fecal Occult Blood Test (FOBT) or fecal immunochemical test (FIT) not completed in the last year
* Complete contact information on file
* Not incarcerated or homeless

Exclusion Criteria:

* Under 50 or over 74 years of age
* Insured but not underinsured
* Other than English or Spanish speaking
* History of colon cancer or colon resection
* History of inflammatory bowel disease
* Colonoscopy completed within the last 10 years
* Sigmoidoscopy completed within the last 5 years
* FOBT or FIT screening completed within the last year
* Incomplete contact information (i.e., no address or phone number on file)
* Incarcerated or homeless

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7711 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Increase in colorectal cancer screening rate of the 5 tested invitation approaches. | 24 days [3 week + 3 days for mailing] from time of mailed invitation
  Primary analysis will be proportion of participants returning their kit within 24 days of mailing. We a priori computed sample size required to have 80% power to detect at least an 8% absolute increase in screening between each branch. We planned for 10 pairwise comparisons with a two-sided 0.005 (=0.05/10) significance level and Bonferroni correction. Estimated return rate for the control was 36.5%. Based on these parameters, we estimate requiring at least 1,026 individuals per group. To maximize sample receiving outreach, the final sample will randomize all eligible patients and is expected to be larger than 1,026 per group.

CONTACTS AND LOCATIONS:
Overall Officials: Keith E Argenbright, MD, Principal Investigator — UT Southwestern Medical Center, Moncrief Cancer Institute; Samir Gupta, MD, Study Director — University of California, San Diego
Locations (2):
- United States (2):
  - John Peter Smith Health Network, Fort Worth, Texas
  - UT Southwestern Medical Center, Moncrief Cancer Institute, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010 Sep-Oct;60(5):277-300. doi: 10.3322/caac.20073. Epub 2010 Jul 7. PMID 20610543
- [Background] StatBite: National Costs for Cancer Care in 2010 in Billions of Dollars by Cancer Site. J Natl Cancer Inst. 2012 Jan 4;104(1):13. doi: 10.1093/jnci/djr534. Epub 2011 Dec 14. No abstract available. PMID 22173584
- [Background] Ward E, Halpern M, Schrag N, Cokkinides V, DeSantis C, Bandi P, Siegel R, Stewart A, Jemal A. Association of insurance with cancer care utilization and outcomes. CA Cancer J Clin. 2008 Jan-Feb;58(1):9-31. doi: 10.3322/CA.2007.0011. Epub 2007 Dec 20. PMID 18096863
- [Background] Hardcastle JD, Chamberlain JO, Robinson MH, Moss SM, Amar SS, Balfour TW, James PD, Mangham CM. Randomised controlled trial of faecal-occult-blood screening for colorectal cancer. Lancet. 1996 Nov 30;348(9040):1472-7. doi: 10.1016/S0140-6736(96)03386-7. PMID 8942775
- [Background] Mandel JS, Bond JH, Church TR, Snover DC, Bradley GM, Schuman LM, Ederer F. Reducing mortality from colorectal cancer by screening for fecal occult blood. Minnesota Colon Cancer Control Study. N Engl J Med. 1993 May 13;328(19):1365-71. doi: 10.1056/NEJM199305133281901. PMID 8474513
- [Background] Kronborg O, Fenger C, Olsen J, Jorgensen OD, Sondergaard O. Randomised study of screening for colorectal cancer with faecal-occult-blood test. Lancet. 1996 Nov 30;348(9040):1467-71. doi: 10.1016/S0140-6736(96)03430-7. PMID 8942774
- [Background] Faivre J, Dancourt V, Lejeune C, Tazi MA, Lamour J, Gerard D, Dassonville F, Bonithon-Kopp C. Reduction in colorectal cancer mortality by fecal occult blood screening in a French controlled study. Gastroenterology. 2004 Jun;126(7):1674-80. doi: 10.1053/j.gastro.2004.02.018. PMID 15188160
- [Background] Atkin WS, Edwards R, Kralj-Hans I, Wooldrage K, Hart AR, Northover JM, Parkin DM, Wardle J, Duffy SW, Cuzick J; UK Flexible Sigmoidoscopy Trial Investigators. Once-only flexible sigmoidoscopy screening in prevention of colorectal cancer: a multicentre randomised controlled trial. Lancet. 2010 May 8;375(9726):1624-33. doi: 10.1016/S0140-6736(10)60551-X. Epub 2010 Apr 27. PMID 20430429
- [Background] Kahi CJ, Imperiale TF, Juliar BE, Rex DK. Effect of screening colonoscopy on colorectal cancer incidence and mortality. Clin Gastroenterol Hepatol. 2009 Jul;7(7):770-5; quiz 711. doi: 10.1016/j.cgh.2008.12.030. Epub 2009 Jan 11. PMID 19268269
- [Background] Brenner H, Chang-Claude J, Seiler CM, Rickert A, Hoffmeister M. Protection from colorectal cancer after colonoscopy: a population-based, case-control study. Ann Intern Med. 2011 Jan 4;154(1):22-30. doi: 10.7326/0003-4819-154-1-201101040-00004. PMID 21200035
- [Background] Baxter NN, Goldwasser MA, Paszat LF, Saskin R, Urbach DR, Rabeneck L. Association of colonoscopy and death from colorectal cancer. Ann Intern Med. 2009 Jan 6;150(1):1-8. doi: 10.7326/0003-4819-150-1-200901060-00306. Epub 2008 Dec 15. PMID 19075198